CLINICAL TRIAL: NCT01572415
Title: Evaluation of SCOUT DS Device in the Diagnosis of Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: VeraLight, Inc. (Industry)
Collaborators: Greece National Social Insurance Institute (Unknown); Laikο General Hospital, Athens (Other)
Responsible Party: Sponsor
Other Study IDs: VL-MK01
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes
Keywords: Screening for Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to identify compare SCOUT DS to random capillary glucose for identification of at-risk subjects with dysglycemia defined by hemoglobin A1C ≥ 6.0%.

DETAILED DESCRIPTION:
The study will complete up to 400 subjects at the clinical site to evaluate the precision and accuracy of SCOUT DS and random capillary glucose for detecting pre-diabetes and undiagnosed type 2 diabetes in subjects at risk but not having a pre-existing diagnosis of type 2 diabetes. A point of care A1c measurement will serve as the reference method for defining pre-diabetes (6.0% ≤ A1c ≤ 6.4%) and diabetes (A1c ≥ 6.5%).

The study will require one visit by each subject to the clinical site. The visit does not require fasting and can be done any time of day. The study (not including the IRB process and recruiting) is expected to last 6 months.

The target cohort for comprises persons at risk for pre-diabetes and/or type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 45 years

OR

Age 18 to 44 years and with one or more of the following risk factors:

* BMI > 25 kg/m²
* Elevated waist circumference, > 35 inches for women and >40 inches for men
* Habitually physically inactive (does not exercise regularly)
* Has a first-degree relative with diabetes
* Ethnicity with elevated risk for type 2 diabetes
* Has delivered a baby weighing > 9 lb or diagnosed with gestational diabetes
* Hypertension (≥130/≥ 85 mmHg) or being treated for hypertension
* HDL cholesterol level < 35 mg/dL and/or a fasting triglyceride level ≥ 250 mg/dL or being treated for dyslipidemia with medication
* Has been previously diagnosed with Polycystic Ovary Syndrome (PCOS)
* Had impaired glucose tolerance or impaired fasting glucose on previous testing within the last 3 yrs
* Conditions associated with insulin resistance such as acanthosis nigricans
* History of vascular disease including heart attack, stroke, angina, coronary heart disease, atherosclerosis, congestive heart failure or peripheral arterial disease

Exclusion Criteria:

* • Under 18 years of age

  * Receiving investigational treatments in the past 14 days
  * Psychosocial issues that interfere with an ability to follow study procedures
  * Conditions that cause secondary diabetes including Cushing's syndrome, acromegaly, hemochromatosis, pancreatitis, or cystic fibrosis
  * Diagnosed with any type of diabetes, including type 1 or 2
  * Taking glucose lowering medications with the exception of metformin
  * Known to be pregnant
  * Receiving dialysis or having known renal compromise
  * Scars, tattoos, rashes or other disruption/discoloration on the left volar forearm.
  * Recent (within past month) or current oral steroid therapy or topical steroids applied to the left forearm; inhaled steroid therapy is not excluded
  * Current chemotherapy, or chemotherapy within the past 12 months
  * Receiving medications that fluoresce*
  * Known to have, or at risk for, photosensitivity reactions ( e.g., sensitive to ultraviolet light, or taking medication known to cause photosensitivity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects must be 18 years of age or greater.
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Comparison of SCOUT DS to Random Capillary Glucose | Up to 6 months
  A point of care A1c measurement will serve as the reference method for defining pre-diabetes (6.0% ≤ A1c ≤ 6.4%) and diabetes (A1c ≥ 6.5%).
  The study will require one visit by each subject to the clinical site. The visit does not require fasting and can be done any time of day. The study (not including the IRB process and recruiting) is expected to last 6 months.
  The target cohort for comprises persons at risk for pre-diabetes and/or type 2 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Tentolouris, MD, Principal Investigator — LAIKO General Hospital/University of Athens
Locations (1):
- Greece National Social Insurance Institute (IKA), Athens, Greece

REFERENCES:
- [Derived] Tentolouris N, Lathouris P, Lontou S, Tzemos K, Maynard J. Screening for HbA1c-defined prediabetes and diabetes in an at-risk greek population: performance comparison of random capillary glucose, the ADA diabetes risk test and skin fluorescence spectroscopy. Diabetes Res Clin Pract. 2013 Apr;100(1):39-45. doi: 10.1016/j.diabres.2013.01.002. Epub 2013 Jan 28. PMID 23369230